CLINICAL TRIAL: NCT00268294
Title: Restoring Sinus Rhythm With Cardiac Resynchronization in Patients With Atrial Fibrillation
Brief Title: Restoring Sinus Rhythm With Cardiac Resynchronization in Patients With Atrial Fibrillation (ReSync AF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 221
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Heart Failure, Atrial Arrhythmia
Keywords: cardiac resynchronization therapy, atrial arrhythmia
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. When there are changes in the heart beat sometimes an implantable heart device is used to control the rate and rhythm of the heart beat. In certain heart failure cases, when the two lower chambers of the heart no longer beat in a coordinated manner, cardiac resynchronization therapy may be prescribed.

People who have a dangerously fast heart beat, or whose heart is at risk of stopping beating, may be in need of an electronic device called an implantable cardioverter defibrillator (ICD).

Atrial tachyarrhythmia (AT) is the name for rapid beats in the upper chambers of the heart. People with AT may experience symptoms such as heart palpitations (a racing or pounding feeling in the chest), shortness of breath, dizziness, fatigue or weakness.

The purpose of this study is to characterize the impact of cardiac resynchronization therapy versus cardiac resynchronization therapy with atrial therapies on the incidence, duration and termination of atrial tachyarrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with atrial fibrillation
* Subjects with a heart beat that is too fast and who have been determined by a doctor to require an implantable cardioverter defibrillator (ICD) i.

Exclusion Criteria:

* Subjects with a natural heart rate less than 30bpm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-05; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To compare the AF burden, frequency and duration of episodes when atrial therapies are ON vs. OFF.

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Huegl, MD, Principal Investigator — Zentralklinik Bad Berka GmbH
Locations (1):
- Zentralklinik Bad Berka GmbH, Bad Berka, Germany